CLINICAL TRIAL: NCT02849236
Title: Analgesic Efficacy of the Pectoral Nerve Block Type 1 for Breast Subpectoral Implant Surgery: A Randomized Controlled Study
Brief Title: PECS I Block for Breast Subpectoral Implant Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015_17; 2016-000157-12 (EudraCT Number)
Record Dates: First submitted 2016-07-19; First posted 2016-07-29 (Estimated); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Pain, Postoperative
Keywords: PECS block,; pectoral block,; breast augmentation
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Placebo Comparator): PECS block performed with Saline solution instead of local anesthetic
  Interventions: Drug: Placebo
- PECS group (Experimental): PECS block performed with Ropivacaine 3.75mg/mL
  Interventions: Drug: Ropivacaine (PECS bloc)

INTERVENTIONS:
Drug: Ropivacaine (PECS bloc) — Ropivacaine 3.75mg/mL
  Injection of a local anesthetic between pectoral major and pectoral minor muscles
  Other Names: ropivacaine
  Arms: PECS group
Drug: Placebo — 20 mL saline 0.9%
  Other Names: saline
  Arms: Control group

SUMMARY:
Breast augmentation surgery can cause important postoperative pain, especially when bilateral subpectoral implants are used. The investigators hypothesized that a technique of regional analgesia, the pectoral nerve block type I (or "PECS I block") would reduce pain within the first twenty-four hours and, in turn, morphine consumption and associated side effects. This is a randomized, controlled, double-blind study which compares intra and postoperative analgesia with or without PECS I block in breast surgery.

ELIGIBILITY:
Inclusion Criteria:

* Every female who will benefit of a bilateral subpectoral breast augmentation
* Age more than 18 years
* Social insured

Exclusion Criteria:

* refusal of the patient
* Age less than 18 years
* Inability to consent
* History of thoracic surgery or breast implants
* Pregnancy
* Inability to use a patient controlled analgesia
* Contraindication of the use of opioids or local anesthetics
* Pathology of hemostasis, infection
* Can not use a PCA
* Patients under long-term opioids (WHO pain ladder 2 and 3)
* Patient presenting neuropathic pain during the preoperative period (score greater than or equal to 4 to the DN4 questionnaire, or taking anti-epileptic or antidepressant treatments for neuropathic pain)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-10-16 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | During the first 24 postoperative hours
  Morphine consumption by use of patient control analgesia within the first twenty-four hours after surgery.

SECONDARY OUTCOMES:
First administration of morphine | During the first 24 postoperative hours
  Time elapsed between tracheal extubation and first administration of morphine
Post-operative nausea and/or vomiting | During the first 24 postoperative hours
  Number of nausea and/or vomiting episodes in the twenty-four hours after surgery
Intra-operative opioids consumption | During procedure execution
  Sufentanil consumption during anesthesia
Post-operative anti-emetic consumption | During the first 24 postoperative hours
  Consumption of anti-emetic drugs after surgery
Post-operative pain | During the first 24 postoperative hours
  Evaluation of post-operative pain with a digital scale from 0 to 10 in the first twenty four hours after surgery
4-point sedation scale | During the first two postoperative hours
  using WHO Sedation scale
  - 0 = awake and alert /- 1 = quietly awake / - 2 = asleep but easily roused / - 3 = deep sleep
Aldrete score | During the first two postoperative hours
  Aldrete Score is a medical scoring system for the measurement of recovery after anesthesia (post anesthesia) which includes activity, respiration, consciousness, blood circulation and color.
Time physiological function recovery | During the first six postoperative hours after tracheal extubation
  Ability to drink, to eat, to urinate, to walk

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Tavernier, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHU de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No